CLINICAL TRIAL: NCT03504618
Title: Research on the Treatment of Metastatic Colon Cancer Patients Treated by FOLFOXIRI Regimen (Folinic Acid, 5-fluorouracil, Oxaliplatin and Irinotecan)
Brief Title: Research on the Treatment of Metastatic Colon Cancer Patients Treated by FOLFOXIRI
Status: Completed | Type: Observational
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Bui My Hanh, Director, Science Research and International Cooperation Unit, Hanoi Medical University
Other Study IDs: HMU16223
Record Dates: First submitted 2018-04-04; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — FOLFOXIRI protocol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic colon cancer patients: Colon cancer patients with metastase at the diagnostic time, impossibility of radical resection, adenocarcinoma, treated by at least 3 cycles of FOLFOXIRI in the first-line in the Oncology and Palliative Care Department
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — Treatment of FOLFOXIRI regimen at first line with dosage:
  Irinotecan: 165 mg / m2, intravenous infusion for 1 hour. Day 1, 15. Oxaliplatin: 85 mg / m2, intravenously for 2 hours Day 1, 15 Calcium folinate 200 mg / m2, intravenously for 2 hours Day 1, 15 5FU 3200 mg / m 2, intravenous infusion continuously for 48 hours Day 1, 2, 3, 15, 16, 17 Every 4 weeks. Each cycle has 2 infusion times, the first one is the first day, the second one is the 15th day

SUMMARY:
Colon cancer with metastase in the diagnose time account for one significant rate and has a increasing trend. The treatment result of this patient group rests modest. The biological therapeutic treatment is still expensive for major part of Vietnamese patients. So that, research on a new affordable and efficacious chemotherapy combination for these patients is extremely necessary in our country The purpose of the study is to comment somes clinico-pathology features of metastatic colon cancer patients whose disease was not radically resectable.

The second aim is to Evaluate the treatment result and toxicity of FOLFOXIRI in these patients

DETAILED DESCRIPTION:
In the world, colorectal cancer is the third most common cancer in male and the second most common cancer in female. In VietNam, the disease is the fourth cancer in male, the sixth cancer in female and increasing recently. About 20-40% of the colon cancer patients had distant metastasis at the time of diagnose, those treatment outcome remains poor (5years survival is about 11%). The targetted therapy medications are still not affordable for majority of Vietnamese patients. So that, 3 cytotoxic drugs (5-Fluoro-Uracil, Oxaliplatin and Irinotecan) remain back-bone in the treatment of metastatic colon cancer.

According to one meta-analysis, the overall survival rate significantly correlated to the use of all 3 these drugs in the treatment time. If patients were give two drugs as the doublet in a line (FOLFOX/XELOX, FOLFIRI/XELIRI), not 100% of patients are treated with all 3 these drugs because some abandonned the following treatment lines. So, the trials that give all 3 drugs in a line (first-line) as triplet (FOLFOXIRI) were carried out and had primirily good outcome. In 2010, FOLFOXIRI were recommended in NCCN guideline.

In VietNam, FOLFOXIRI has been applied to treat patient since 2013. However, since then there was no clinical trial to evaluate the efficacy and the toxicity of this combination. Therefore, we carried out the work "Research on the treatment of metastatic colon cancer patients treated by FOLFOXIRI"

ELIGIBILITY:
Inclusion Criteria:

* 39 colon cancer patients with metastase at the diagnotic time, impossiblity of radical resection, adenocarcinoma, treated by at least 3 cylces of FOLFOXIRI in the first-line in the Oncology and Palliative Care Department, Ha Noi medical university hospital, from September 2013 to April 2017

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited to the study will be explained in detail will be required to sign a volunteer card. All detailed information on the patient's medical condition is encrypted and confidential. The patient has the right to withdraw from the study
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Patients' characteristic | 4 years
  Clinico-pathology features of metastatic colon cancer patients whose disease was not radically resectable
Response rate after 3 cycles | At the end of Cycle 3 (each cycle is 4 weeks)
  Responses are evaluated according to WHO criteria. The determination of responses and progression was initially based on investigator-reported measurements; computed tomography scans of all responding patients and of patients with stable disease were subsequently subjected to external review by an independent panel.
Response rate after 6 cycles | At the end of Cycle 6 (each cycle is 4 weeks)
  Responses are evaluated according to WHO criteria. The determination of responses and progression was initially based on investigator-reported measurements; computed tomography scans of all responding patients and of patients with stable disease were subsequently subjected to external review by an independent panel.
Correlation between response rate and percentage of chemotherapy dosage | 4 years
  Prognostic factor of response rate
Correlation between response rate and histopathology | 4 year
  Prognostic factor of response rate
Correlation between response rate and metastatic site | 4 years
  The average size of the hepatic metastatic lesion in the study
Prognostic factor for response rate after 3 cycles | At the end of cycle 3 (each cycle is 4 weeks)
  Evaluation of predictor of response rate
Prognostic factor for response rate after 6 cycles | At the end of cycle 6 (each cycle is 4 weeks)
  Evaluation of predictor of response rate
Mean of the progression free survival | 4 years
  The median progression free survival of the study population
Prognostic factor of progression free survival | 4 years
  Evaluation of predictor of progression free survival

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 4 years
  During the full length of first-line treatment, number of enrolled patients reporting adverse events is recorded. Adverse events are evaluated according to National Cancer Institute Common Toxicity Criteria latest version.
Overall survival after 12 months | 12 months after the last patient finish chemotherapy
  The percentage of survival patients 12 month after finishing treatment with FOLFOXIRI regimen
Overall survival after 24 months | 24 months after the last patient finish chemotherapy
  The percentage of survival patients 24 month after finishing treatment with FOLFOXIRI regimen

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code